CLINICAL TRIAL: NCT02112162
Title: Pilot Study of Gene Expression and FDG-PET/MR Biomarkers for Evaluation of Response to Neoadjuvant Therapy for Locally Advanced Rectal Cancer
Brief Title: Gene Expression and FDG PET/MRI in Evaluating Treatment Response in Patients With Locally Advanced Rectal Cancer Undergoing Chemotherapy and Radiation Therapy Before Surgery
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Loss of funding
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201401064
Record Dates: First submitted 2014-04-09; First posted 2014-04-11 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Rectal Neoplasms
MeSH Terms: conditions — Rectal Neoplasms | interventions — Fluorodeoxyglucose F18; Positron-Emission Tomography; Tomography; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diagnostic (FDG PET/MRI, gene expression) (Experimental): FDG PET/MRI at baseline and at 2-4 weeks before surgery (after neoadjuvant chemoradiation). Tissue samples for gene expression at baseline and during surgery
  Interventions: Radiation: fludeoxyglucose F 18; Device: positron emission tomography; Device: magnetic resonance imaging; Other: laboratory biomarker analysis

INTERVENTIONS:
Radiation: fludeoxyglucose F 18 — Undergo FDG PET/MRI
  Other Names: 18 FDG, 18FDG, 2-F18-fluoro-2-deoxy-D-glucose, 2-F18-fluoro-2-deoxyglucose, 63503-12-8, FDG, Fluorine-18 2-Fluoro-2-deoxy-D-Glucose, Fluorodeoxyglucose F18
Device: positron emission tomography — Undergo FDG PET/MRI
  Other Names: FDG-PET, PET, PET scan, tomography, emission computed
Device: magnetic resonance imaging — Undergo FDG PET/MRI
  Other Names: MRI, NMR imaging, NMRI, nuclear magnetic resonance imaging
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies gene expression analysis and fludeoxyglucose F 18 (FDG) positron emission tomography (PET)/magnetic resonance imaging (MRI) in evaluating treatment response in patients with rectal cancer that has spread to nearby tissue or lymph nodes undergoing chemotherapy and radiation therapy before surgery. Studying samples of tissue in the laboratory may help doctors learn more about changes that occur in deoxyribonucleic acid (DNA) and may also help doctors predict a patient's response to treatment before surgery. PET-MRI is a procedure that combines the pictures from a PET scan and an MRI scan. The combined scans give more detailed pictures of areas inside the body than either scan gives by itself. PET-MRI may help determine how well people respond to pre-surgery chemotherapy and radiation therapy and help the surgeon make the best plan for removal of the tumor.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven adenocarcinoma of the rectum.
* Surgical candidate.
* Candidate for neoadjuvant chemotherapy.
* Clinical evidence of T1-3N1 or T3N0 disease. This can be either by imaging studies or by physical exam findings.
* At least 18 years of age.
* Zubrod performance status of 0-2.
* Able to understand and willing to sign a written informed consent document.
* Patients with distant metastatic disease will be eligible if they satisfy all other conditions.

Exclusion Criteria:

* Pregnant.
* Past history of pelvic radiotherapy.
* Received prior chemotherapy for colorectal cancer.
* Uncontrolled diabetes with a fasting glucose ≥ 200 mg/dl at the time of PET/MRI imaging.
* Claustrophobia or any other contraindication to MRI imaging evaluated by a standardized safety questionnaire.
* Renal insufficiency (defined as glomerular filtration rate (GFR < 30 mL/min/1.73 m2) measured no more than 60 days before the first research scan) which precludes safe administration of the contrast agent.
* Currently on dialysis.
* Known prior allergic reaction to gadolinium-based MR contrast agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-06; Primary Completion 2015-03 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in FDG-PET/MR SUVmax | Baseline to up to 2 weeks before surgery
  Images will be evaluated semi-quantitatively. Changes in imaging parameters will be correlated with pathologic response.
Change in FDG-PET/MR SUVmean | Baseline to up to 2 weeks before surgery
  Images will be evaluated semi-quantitatively. Changes in imaging parameters will be correlated with pathologic response.
Change in ADCmean | Baseline to up to 2 weeks before surgery
  Images will be evaluated semi-quantitatively. Changes in imaging parameters will be correlated with pathologic response.
Radiosensitivity index | Baseline
  Index is calculated based on tumor gene expression. Will be correlated with the descriptive changes in FDG-PET/MR SUV and ADC parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Parag Parikh, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu